CLINICAL TRIAL: NCT02284672
Title: The Effect of Dexmedetomidine on Propofol Requirement for Insertion of Laryngeal Mask Airway
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, clinical assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AJIRB-MED-CT4-14-296
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Precedex Effect to Propofol Requirement
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): After preoxygenation for 3 minutes, normal saline would be injected to patient for 10 minute. First, 1% lidocaine 3 ml were given for reducing injection pain of propofol and the settled amount of propofol was injected during 15 seconds.
  After 90 seconds, other anesthesiologist who did'nt know the injected drug tried to insert LMA.
  Interventions: Drug: Normal saline
- dexmedetomidine (Experimental): After preoxygenation for 3 minutes, dexmedetomidine would be injected to patient for 10 minute. First, 1% lidocaine 3 ml were given for reducing injection pain of propofol and the settled amount of propofol was injected during 15 seconds.
  After 90 seconds, other anesthesiologist who did'nt know the injected drug tried to insert LMA.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: dexmedetomidine
Drug: Normal saline
  Arms: control

SUMMARY:
Propofol frequently used as an inducting medication for insertion Laryngeal mask airway(LMA). But propofol alone can be not sufficient for inhibiting upper airway reflex and also result in cardiovascular suppression under enough amount. Dexmedetomidine is a selective alplh2 receptor agonist with analgesic and sedative effects but sparing respiratory function. Therefore propofol combined with dexmedetomidine induction could be more effective in preserve respiration under same condition for LMA insertion than propofol alone. In this study, the investigators investigate the clinical dose of propofol for LMA insertion with premedication of dexmedetomidine, and evaluate the effect of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* patients for surgery not exceed more than 2 hours requiring general anesthesia

Exclusion Criteria:

* history of gastroesophageal reflux High grade obesity Predicted diffiicult airway

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Fail or success for Laryngeal Mask Airway (LMA) insertion | During inserting LMA and up to 5 seconds after LMA inserion
  Failure for LMA insertion is defined if there is a difficulty for mouth opening or active movement of four limbs or head. Success is smooth LMA insertion without any movement

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Yoo, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Jiyoung Yoo, Suweon, Kyunggido, South Korea